CLINICAL TRIAL: NCT06104228
Title: 129 Xenon MRI as a Biomarker for Diagnosis and Response to Therapy in Pulmonary Arterial Hypertension (PAH)
Acronym: Xenon PAH Bio
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bastiaan Driehuys (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Bastiaan Driehuys, Professor of Radiology, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00113893
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Arterial Hypertension; Pulmonary Arterial Hypertension Associated With Connective Tissue Disease (Disorder); Connective Tissue Diseases
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Idiopathic Pulmonary Arterial Hypertension (Other): Arm 1... patients with IPAH
  Interventions: Drug: 129Xe Hyperpolarized
- Pulmonary Arterial Hypertension Associated with Connective Tissue Disease (Other): Arm 2... patients with CTD-PAH
  Interventions: Drug: 129Xe Hyperpolarized

INTERVENTIONS:
Drug: 129Xe Hyperpolarized — Each xenon dose will be limited to a volume less than 25% of a subject's total lung capacity (TLC), as is the case for all protocols currently carried out under IND 109490

SUMMARY:
The overall study objectives outlined in this study are to derive 129Xe MRI pulmonary vascular biomarker signatures that differentiate common subtypes of PAH and to determine the ability of 129Xe MRI to longitudinally monitor disease progression and response to therapy in PAH, with the aid of additional assessments, such as labs, echocardiography, and six-minute walk distance (6MWD).

DETAILED DESCRIPTION:
Subject Enrollment This study will consent and enroll 20 subjects total.

• For Arm 1, 10 subjects with Idiopathic Pulmonary Arterial Hypertension (IPAH) will be consented and enrolled. For Arm 2, 10 subjects with Connective Tissue Disease Associated Pulmonary Arterial Hypertension (PAH-CTD) will be consented and enrolled.

Study Design This study will be observational. Subjects in both arms of the trial will undergo a 129Xe MRI/MRS at timepoints of baseline, 3 months, 6 months, and 12 months. In addition to the this, data from standard of care assessments, such as labs, echocardiography, and six-minute walk distance (6MWD), will also collected at these timepoints.

Primary Study Endpoints The primary endpoint for this trial will be the change in defect + low percentage of RBC signal on hyperpolarized 129Xe MRI from baseline to 12 months

Secondary Study Endpoints

There will be several secondary endpoints for this trial:

* Change in regional and global RBC Oscillation Amplitudes on hyperpolarized 129Xe MR spectroscopy from baseline to 12 months
* Change in 6MWD from baseline to 12 months
* Change in NTproBNP from baseline to 12 months
* Change in WHO FC from baseline to 12 months

Primary Safety Endpoints

There will be several primary safety endpoints for this trial:

* Frequency of Adverse Events (AE) and/or Serious Adverse Events (SAE)
* Withdrawals due to adverse event or death
* Incidence of Adverse Events of Significant Interest (AESI):
* Electrocardiogram and any findings
* Physical examination and vital signs

ELIGIBILITY:
Inclusion Criteria:

Arm 1 -IPAH

* Age: 18-75 years
* WHO functional class 2 or 3
* Mean pulmonary artery pressures > 20 mmHg
* Pulmonary capillary wedge pressure ≤15 mmHg
* Pulmonary vascular resistance > 2 Wood Units (WU)
* No other cause identified for PAH

Arm 2 -PAH-CTD

* Age: 18-75 years
* WHO functional class (FC) 2 or 3
* Mean pulmonary artery pressures > 20 mmHg
* Pulmonary capillary wedge pressure ≤15 mmHg
* Pulmonary vascular resistance > 2 WU
* Diagnosis of connective tissue disease

Exclusion Criteria:

* PH other than Idiopathic PAH or PAH associated with CTD; any conditions that prevent the performance of 129Xe MRI scans will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Remodeling | 1 year
  The primary endpoint for this trial will be the change in defect + low percentage of RBC signal on hyperpolarized 129Xe MRI from baseline to 12 months

SECONDARY OUTCOMES:
RBC Oscillation Amplitude | 1 year
  • Change in regional and global RBC Oscillation Amplitudes on hyperpolarized 129Xe MR spectroscopy from baseline to 12 months
6 Minute Walk Distance | 1 Year
  Change in 6MWD from baseline to month 12
NTproBNP | 1 year
  Change in NTproBNP from baseline to month 12
World Health Organization (WHO) Functional Class (FC) | 1 year
  Change in WHO FC from baseline to month 12

CONTACTS AND LOCATIONS:
Overall Officials: Fawaz Alenezi, MD, Principal Investigator — Duke Univeristy
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No